CLINICAL TRIAL: NCT04842214
Title: Evaluation of Disease Course in Oncological Patients During Inpatient Rehabilitation and After Three Months Follow-up: a Cohort Study.
Brief Title: Disease Course in Oncological Patients During Inpatient Rehabilitation and After Three Months Follow-up
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Klinik Valens (Other)
Responsible Party: Principal Investigator, Jens Bansi, Head of Research and Development, Klinik Valens
Other Study IDs: Bansi-2021
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Oncologic Disorders
Keywords: Oncologic Rehabilitation; Cancer-related Fatigue; Patient-reported Outcome Measurement Information System (PROMIS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Oncologic disorders: All patients assigned for oncological rehabilitation with the diagnosis "Cancer" are included to this cohort.
  Interventions: Behavioral: Oncological Rehabilitation

INTERVENTIONS:
Behavioral: Oncological Rehabilitation — Multidimensional rehabilitation

SUMMARY:
Constant improvements in the areas of diagnostics and treatment lead to an increase of patients surviving an oncological diagnosis ("cancer survivors") thus increasing the cost factor on both society and health care systems. Meta-analysis have shown the effectiveness of multidimensional rehabilitation programs concerning cost-effectiveness and for improving different health parameters. However when submitted to oncological rehabilitation in Switzerland there is no clear definition when to use which specific assessment during the different stages of oncological rehabilitation.

This cohort study aims to evaluate and systematically follow-up patients that are assigned for oncological inpatient rehabilitation at the Rehabilitation Center Walenstadtberg.

The main purposes are i) to evaluate disease onset of oncological patients during rehabilitation and to identify relationships between mobility and cancer-related fatigue at discharge; ii) to identify predictive factors for everyday functioning and social participation after three months discharge.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with "Cancer";
* Literacy and understanding German language;
* Signed informed consent;

Exclusion Criteria:

* Women who are pregnant or breastfeeding / have the intention to become pregnant during the course of the study;
* Other clinically significant concomitant disease states (e.g. renal failure, hepatic dysfunction, cardiovascular disease, etc);
* Known or suspected non-compliance, drug or alcohol abuse;
* Inability to follow the procedures of the study: e.g. due to language problems, psychological disorders, dementia of the participant, etc;
* Enrolment of the investigator, his/her family members, employees and other dependent persons;
* Cognitive impairment: Mini-Mental State Examination (MMSE) < 21;
* Major Depression or Hospital Anxiety and Depression Scale (HADS) >11 at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with oncologic disorders assigned for inpatient rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) | Three months (Day 0-Day 92) with time points set after three weeks (Day 21) and three months (Day 92)
  Change of participants' physical and mental health over three weeks training and after three months discharge (follow-up). The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score with higher scores indication better physical and/or mental health.

SECONDARY OUTCOMES:
Multidimensional Fatigue Inventory (MFI) | Three months (Day 0 - Day 92) with time points set after three weeks (Day 21) and three months after discharge (Day 92)
  Changes of cancer-related fatigue over three training weeks and after three months follow-up. The MFI is a 20-item self-report instrument designed to measure fatigue. It covers the following dimensions: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. The scale ranges from 1 to 7 with higher total scores indicating acute levels of fatigue.
Functional Independence Measure (FIM) | Three weeks (Day 0 - Day 21)
  Changes of participants functional independencies of performing a task over three weeks training. The FIM is a 18-item self-report instrument designed to measure participants functional independency. Items are divided into motor and cognitive categories, are classified based on the type of task it involves and are scored on a 7-point likert scale. Higher scores indicate more independencies a person has at performing the task. The score is a value ranging between 18 and 126 (total score) and is further broken down based on its motor and cognitive components. The motor component ranges from 13 to 91, while the cognitive component ranges between 5 to 35.
EuroQoL-Group five dimension quality of life questionnaire (EQ-5D) | Three weeks (Day 0 - Day 21)
  Changes of participant's health state over three weeks training with higher scores indicating a better health status.EQ-5D comprises the five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is expressed with the levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by scoring the most appropriate statement for each dimension. This decision results into a 1-digit number that expresses the level selected for the respective dimension. The digits for the five dimensions are combined into a 5-digit number.
Six Minute Walking Test (6MWT) | Three weeks (Day 0 - Day 21)
  Changes of walking speed and distance covered after in 6-Minutes over three weeks training. The greater the distance covered after six minutes the higher the walking speed.
Timed-Up-and-Go (TUG) | Three weeks (Day 0 - Day 21)
  Changes of mobility and risk of falling over three weeks training. The TUG measures the time for the participant to stand from a chair, walk three meters and sit down again. Time stops when the participants is seated. Cut-off for risk of falling is set for dwelling adults at 13.5 and for vestibular disorders at 11.1 seconds.
Hospital Anxiety and Depression Scale (HADS) | Three weeks (Day 0 - Day 21)
  Changes of anxiety and depression over three weeks training on a 4-point likert scale scored 0-3. Max 21 Points for each subscale, cut off for anxiety and Depression are set at 7 points with higher values representing more anxiety and depressive symptoms symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Kliniken-Valens, Valens, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No